CLINICAL TRIAL: NCT02758379
Title: Early Safety and Feasibility Study of the Shockwave Coronary Lithoplasty™ System in Coronary Arteries
Brief Title: Shockwave Coronary Lithoplasty Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Collaborators: Yale Cardiovascular Research Group (Other); Massachusetts General Hospital (Other); Pacific Clinical Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD 0200
Record Dates: First submitted 2015-01-16; First posted 2016-05-02 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Coronary Stenosis
Keywords: coronary artery disease; calcified lesions; lithotripsy
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Shockwave Coronary Lithoplasty System (Experimental): Patients receive Lithoplasty treatment prior to placement of coronary stent. IVUS or OCT documents patency pre and post Lithoplasty. Patient is followed for patency at discharge, 30 days and 6 months following treatment.
  Interventions: Device: Shockwave Coronary Lithoplasty System

INTERVENTIONS:
Device: Shockwave Coronary Lithoplasty System — Lithotripsy shockwaves are used to fracture calcified lesions in the coronary arteries

SUMMARY:
The objective of this clinical trial is to study the early safety and feasibility of the Shockwave Coronary Lithoplasty System. To demonstrate that the Shockwave device can safely and effectively deliver localized shockwave energy for balloon dilatation of calcified, stenotic, de novo coronary lesions.

DETAILED DESCRIPTION:
Prospective, non-randomized, single center First In Human (FIH) trial for treatment of stenotic calcified coronary lesions with the Shockwave Lithoplasty System. Patients will be enrolled and consented in the study based on history and in some instances an angiogram obtained prior to the study. The study is designed to demonstrate that the Shockwave device can safely and effectively deliver localized shockwave energy for balloon dilatation of calcified, stenotic, coronary arteries. Subjects will be prepared for PCI per the institution's standard protocol. Medications will be administered per the treatment protocol. Femoral access will be obtained using a 6F access sheath, and guiding catheter placed at the ostia of the right or left coronary artery. Baseline angiography of the culprit lesion will be performed prior to placement of a 0.014" guide wire. Baseline and either IVUS or OCT will be performed to determine the Maximum Lumen Area (MLA), percent stenosis, and volumetric lesion assessment. Baseline angiography will be performed to determine lesion length, % stenosis and reference vessel diameter. The investigational device will be prepped per the IFU and positioned at the target lesion. The distal end of the balloon catheter will be connected to the patient cable. The balloon catheter will be inflated to 4 atm and the investigator will deliver 10 pulses for 20 seconds. The balloon will then be inflated to reference vessel diameter and then deflated to reestablish flow and complete one treatment cycle. The treatment cycle will then be repeated. Angiography and either IVUS or OCT will be repeated for the treated lesion.. A coronary stent will be deployed at the site of treatment. Angiography and either IVUS or OCT will be performed following stent placement. Patients will be followed through discharge and at 30 and 180 days. A subset of up to five (5) subjects will receive an angiographic assessment at the 180 day follow up visit, per the Sponsor's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age and able to give informed consent.
2. Patients in Sinus Rhythm.
3. Patients with significant (> 50% diameter stenosis) native coronary artery disease including stable or unstable angina and silent ischemia, suitable for PCI.
4. Ability to tolerate dual antiplatelet agent (i.e. aspirin, clopidogrel or prasugrel). For 1 year and single therapy for life.
5. Patient is able and willing to comply with all assessments in the study.
6. Stenosis of LAD, RCA or LCX artery ≥50% in a reference vessel of 2.5mm-3.5 mm diameter and ≤ 22 mm length, as assessed by two orthogonal angiographic views.
7. Calcification with parallel calcium at least 50% the length of the lesion.
8. At the time of the procedure the subject is in Sinus Rhythm.
9. Single lesions per vessel.
10. Ability to pass a 0.014" guide wire across the lesion.

Exclusion Criteria:

1. Concomitant use of Rotablator, Cutting Balloon, or investigational coronary devices.
2. Additional planned coronary interventions for a non-target lesion within 180 days of the study procedure.
3. Left ventricular ejection fraction < 40%
4. Patients refusing or not candidates for emergency coronary artery bypass grafting (CABG) surgery
5. Uncontrolled severe hypertension (systolic BP >180 mm Hg or diastolic BP >110 mm Hg)
6. Patients who are not candidates for dual anti-platelet therapy for 30 days and chronic single anti-platelet therapy
7. Severe renal failure with creatinine >2.5 mg/dL
8. Untreated pre-procedural hemoglobin <10 g/dL
9. Coagulopathy manifested by platelet count <100,000 or International Normalized ratio (INR) >1.7 (INR is only required in patients who have taken warfarin within 2 weeks of enrollment)
10. Patients in cardiogenic shock
11. Acute myocardial infarction (MI) within the past one (1) month, and/or elevated CPK (and abnormal Troponin-I) at the time of enrollment
12. Patients with a life expectancy of less than 1 year
13. Target main branch vessel < 2.5 mm in diameter
14. Target main branch lesion > 22 mm in length
15. Chronic Total Occlusion (CTO).
16. Previous stent procedure within 10 mm of target lesion
17. Prior PCI procedure within the last 6 months.
18. Target lesion demonstrating severe dissection prior to planned use of the Shockwave device
19. Unprotected Left Main diameter stenosis ≥ 50%
20. Visible thrombus (by angiography) at target lesion site
21. Patient has active systemic infection
22. Patient with an externally-connected intracardiac catheter or pacemaker.
23. Patient with an implantable pacemaker or defibrillator.
24. Patient has connective tissue disease (e.g., Marfan's syndrome)
25. Patient has a hypercoagulable disorder.
26. Patient has allergy to imaging contrast media for which they cannot be pre-medicated.
27. Evidence of aneurysm or acute thrombus in target vessel.
28. Patients with prior sternotomy as a result of thoracic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Safety - Acute, as indicated by number of subjects that do not experience death following delivery of shockwave energy | Post-procedure (within 24 hours following procedure)
Safety - Acute, as indicated by number of subjects that do not experience tamponade following delivery of shockwave energy | Post-procedure (within 24 hours following procedure)
Safety - Acute, as indicated by number of subjects that do not experience dissection, occlusion or perforation of the coronary artery that requires additional intervention to treat besides stenting following delivery of shockwave energy | Post-procedure (within 24 hours following procedure)
Safety - Acute, as indicated by number of subjects that do not experience aneurysm following delivery of shockwave energy | Post-procedure (within 24 hours following procedure)
Safety - Acute, as indicated by number of subjects that do not experience MI (CPK > 5 x uln) following delivery of shockwave energy | Post-procedure (within 24 hours following procedure)
Safety - Acute, as indicated by number of subjects that do not experience cardiogenic shock following delivery of shockwave energy | Post-procedure (within 24 hours following procedure)
Safety - Acute, as indicated by number of subjects that do not experience distal embolization compromising blood flow, and requiring intervention following delivery of shockwave energy | Post-procedure (within 24 hours following procedure)
Safety - Acute, as indicated by number of subjects that do not experience blood transfusion due to excessive blood loss following delivery of shockwave energy | Post-procedure (within 24 hours following procedure)
Safety - Acute, as indicated by number of subjects that do not experience stroke following delivery of shockwave energy | Post-procedure (within 24 hours following procedure)
Safety - 30 days (Number of subjects without any procedure and/or device related adverse events) | 30 days post procedure
Safety - 30 days (Number of subjects without target lesion revascularization (TLR) | 30 days post procedure
Safety - 30 days (Number of subjects without groin complications) | 30 days post procedure
Safety - 180 days (Number of subjects without any procedure and/or device related adverse events) | 180 days post procedure
Safety - 180 days (Number of subjects without any target lesion revascularization (TLR)) | 180 days post procedure
Performance - Acute technical success of the device | Post-procedure (within 24 hours following procedure)
  * Successful delivery of the device and administration of lithotripsy-enhanced low pressure balloon dilation to the target lesion
  * Residual stenosis of ≤50% of the reference vessel size of the target lesion assessed by angiography and either IVUS or OCT.
  * Successful access of the treatment site with a coronary stent
Safety - Acute, as indicated by number of subjects that do not experience ventricular arrhythmic event requiring intervention to re-establish normal rhythm following delivery of shockwave energy | Post-procedure (within 24 hours following procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Whitbourn, M.D., Principal Investigator — St. Vincent Hospital, Melbourne, Australia
Locations (1):
- St. Vincent's Hospital Melbourne, Melbourne, Victoria, Australia